CLINICAL TRIAL: NCT03337971
Title: Evaluation of a Milk-Based Nutritional Supplement to Modify Diurnal Rates of Bone Turnover and Effect a Positive Change in Bone Health in Post-Menopausal Women at Risk of Osteoporosis
Brief Title: Nutritional Supplement and Bone Health in Post-Menopausal Women
Acronym: MBPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Dairygold Cooperative Society Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IP2016_0476; IP2016_0476 (Other Grant/Funding Number: Enterprise Ireland)
Record Dates: First submitted 2017-10-12; First posted 2017-11-09 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Bone and Bones; Osteoporosis Risk; Osteoporosis, Postmenopausal
Keywords: Post-menopausal; Osteoporosis; Bone Turnover Markers; Dairy Products
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: A block randomised, cross-over design receiving either a milk-based protein supplement (MBPS) or isoenergetic (corn starch) placebo control (PLACEBO).
Who Masked: Participant
Masking Description: Single blind (participant only)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLACEBO (Placebo Comparator): Intervention: Dietary Supplement: PLACEBO A group of subjects ingesting a liquid beverage (0.3g per kg body mass ; 1.2kcal/kg body mass) at 10:00pm, 3h post-absorptive of a standardised evening meal.
  Samples for the measurement of biomarkers of change in the rate of bone turnover appearing in the blood to be collected for the immediate 4h, and excreted in urine, 24h post-ingestion
  Interventions: Dietary Supplement: PLACEBO
- Milk-based protein matrix (Active Comparator): Intervention: Dietary Supplement: MBPM A group of subjects ingesting a liquid beverage (0.3g per kg body mass ; 1.2kcal/kg body mass) at 10:00pm, 3h post-absorptive of a standardised evening meal.
  Samples for the measurement of biomarkers of change in the rate of bone turnover appearing in the blood to be collected for the immediate 4h, and excreted in urine, 24h post-ingestion
  Interventions: Dietary Supplement: MBPM

INTERVENTIONS:
Dietary Supplement: PLACEBO — A food-grade proprietary product containing corn starch in powder form, flavoured and instantised to be dissolved in water. Supplied by Dairygold Ingredients, Mitchelstown, Co Cork, Ireland
  Arms: PLACEBO
Dietary Supplement: MBPM — A food-grade proprietary product containing per 100g; milk protein (46.4%), carbohydrate (40.6%), fat (0.7%), Vitamin D (2ug); calcium (1840mg) in powder form, flavoured and instantised to be dissolved in water. Supplied by Dairygold Ingredients, Mitchelstown, Co Cork, Ireland
  Arms: Milk-based protein matrix

SUMMARY:
The process of bone remodeling exhibits pronounced diurnal pattern that is important for bone health. A balanced rate of bone resorption is required to maintain bone health, a balance that can be disturbed during the lifecycle to effect net rate of formation (as occurs during growth and development to adulthood) or net resorption (as occurs, for example, during the menopause).The research to be undertaken investigates the pluripotent effect of dairy-based products on the regulation of the diurnal process of bone metabolism in post-menopausal women at risk of osteoporosis.

DETAILED DESCRIPTION:
Study Design: A block randomised, cross-over design of 24h rates of bone turnover in healthy, post-menopausal women with osteopenia receiving either a milk-based protein supplement (MBPS) or isoenergetic placebo control (PLACEBO).

Participants: 16 Post-menopausal women with osteopenia as determined by site-specific bone mineral density BMD (DXA) diagnosed and screened by a clinician and for dietary intake of calcium and Vit D by a clinical dietitian.

Subject screening (clinical examination) and dietary intake of calcium and Vit D (by food frequency questionnaire) will precede the experimental protocol.

Experimental protocol and data collection:

Subjects will attend for a 2 day and 2 night (overnight) residence equipped to conduct residential human trials.

The subjects' programmed protocol is as follows;

1. Arrive @ 17:00h with overnight bag;
2. Empty bladder and then provide and retain urine samples for the duration of the stay (assisted collection by researchers);
3. Consume a standardised evening meal (pre-prepared by the research dietitian) and then relax reading/watching films etc;
4. At 20:00h a research nurse will insert a cannula into a superficial arm vein and a blood draw (5ml) will be taken and processed for later analysis;
5. Further blood draws (5ml) will be taken at 22:00h, 2300h, 2400h,0100h and 0200h and the cannula withdrawn;
6. At 22:00h consume either placebo control (PLACEBO) (day 1) OR supplement (MBPM)(day 2) - or vice versa - in randomised order.
7. Retire to bedroom;
8. Consume a standardised breakfast and lunch (pre-prepared by the research dietitian) whilst living in and around the University grounds (i.e. in close proximity to ensure 24h urine collection is complete);
9. Repeat from 2 above to end of 2nd day.

ELIGIBILITY:
Inclusion Criteria:

Post-menopausal women aged 50-70y. Assessed by site-specific BMD to be osteopenic. Assessed by clinical screen to be otherwise healthy and free from other illness or current medication likely to influence the study outcome.

Exclusion Criteria:

Intolerance to dairy-based food products

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Bone turnover | Pre-ingestion and1,2,3 and 4hours post-ingestion (serum) and Pre-ingestion to +24hour post-ingestion (urine)
  A balance of the difference between the magnitude and time course of the acute change (0-4h) in serum C-terminal telopeptide of type 1 collagen (CTX) in ng/mL, a measure of bone resorption, and procollagen type 1 amino-terminal propeptide (P1NP) in ng/ml, a measure of bone formation and diurnal change in bone resorption measured by 24h urinary excretion of deoxypyridinoline (Dpd), a marker of bone resorption, normalised to creatinine. Units nmolDPD/mmolCr

SECONDARY OUTCOMES:
Change in regulator of bone metabolism - PTH | Pre-ingestion,1,2,3 and 4hours post-ingestion
  The magnitude and time course of the acute change (0-4h) in serum parathyroid hormone (PTH) measured in pmol/L
Change in regulator of bone metabolism - RANKL | Pre-ingestion,1,2,3 and 4hours post-ingestion
  The magnitude and time course of the acute change (0-4h) in serum receptor activator of the nuclear factor κB ligand (RANKL) measured in ng/dL
Change in regulator of bone metabolism - OPG | Pre-ingestion,1,2,3 and 4hours post-ingestion
  The magnitude and time course of the acute change (0-4h) in serum receptor activator of the osteoprotegerin (OPG) measured in pg/mL
Incretin peptide (GIP) | Pre-ingestion,1,2,3 and 4hours post-ingestion
  The magnitude and time course of the acute change (0-4h) in enterogastric peptide glucose-dependent insulinotropic peptide (GIP1-42) measured in pg/mL
Incretin peptide (GLP-1) | Pre-ingestion,1,2,3 and 4hours post-ingestion
  The magnitude and time course of the acute change (0-4h) in enterogastric glucagon-like peptide-1 (GLP-17-36) measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Co Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Inreventions in Inflammation Infection and Immunity — http://ul.ie/4i

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03337971/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03337971/SAP_000.pdf